CLINICAL TRIAL: NCT06295861
Title: Prospective Cohort Study of Panvascular Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1194
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: ASCVD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASCVD cohort: The patient had atherosclerosis in 2 or more vessels
  Interventions: Other: no different intervention between the two cohort.
- healthy cohort: The patient had no atherosclerosis in vessels
  Interventions: Other: no different intervention between the two cohort.

INTERVENTIONS:
Other: no different intervention between the two cohort. — no different intervention between the two cohort.

SUMMARY:
To construct a comprehensive big data platform for Chinese people with panvascular disease, and establish a Chinese panvascular disease oriented to guide treatment decisions Cohort and imaging, biological database; According to the clinical features, morphological structure, pathological characteristics of panvascularization, vascular age As the core of the evaluation, a standard evaluation system and a risk prediction model of intervention technology suitable for the diagnosis and treatment of patients with panvascular disease in China were established. Into the Further optimize the treatment strategies, protocols and clinical pathways for panvascular disease to improve patient prognosis and promote its application.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old 2. Patients with panvascular disease: i.e., 2 or more of the following vascular diseases.

2.1 Coronary artery: 2.1.1 Coronary atherosclerotic heart disease: including acute coronary syndrome, stable angina, moderate or more stenosis of the coronary artery, history of myocardial infarction, history of coronary revascularization such as stent implantation or bypass grafting.

2.2. Cerebrovascular: 2.2.1 Intracranial atherosclerotic disease: including ischemic stroke, transient ischemic attack or moderate or more stenosis of the intracranial artery.

2.2.2 Cervical atherosclerotic disease: including carotid artery disease, vertebral artery disease.

2.3. Aorta: 2.3.1 Aortic atherosclerotic disease: including severe aortic plaque, aortic ulcer, aortic stenosis or atresia, aortic dissection, aortic aneurysm, etc.

2.4. Peripheral arteries: 2.4.1 Upper limb atherosclerotic disease: including subclavian artery, axillary artery, brachial artery and other sites.

Edition 2 January 25, 2024 2.4.2 Renal atherosclerotic disease 2.4.3 Mesenteric atherosclerotic disease 2.4.4 Lower limb atherosclerotic disease 3. Clinical data and biological samples are available 4. The subjects or their legal representatives were informed of the nature of the study and agreed to all terms of participation in the study, and signed the informed consent approved by the ethics committee of each clinical center.

Exclusion Criteria:

* 1. Currently undergoing treatment for malignant tumor (radiotherapy, chemotherapy, during surgery, etc.) 2. Current medical conditions requiring urgent treatment (this criterion is not excluded after the condition is stabilized): such as acute infection, hypertension crisis, diabetic ketoacidosis, aortic dissection, etc.

  3. Current severe heart failure (NYHA class 4) 4. Current liver failure (ALT or AST ≥ 5 times the upper limit of normal) or current renal failure (decreased renal function caused by any reason (defined as eGFR < 30mL/(min·1.73m2)) 5. Pregnant or lactating women, or women who plan to become pregnant during the study period 6. Current severe mental illness (except mild to moderate anxiety and depression) 7. Organ transplantation 8. Estimated survival time <3 years 9. Blood-borne infectious diseases: including HIV infection, AIDS, active hepatitis B, hepatitis C, etc.

  10. Any condition considered inappropriate for participation in the study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study with 50,000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular adverse events | 1, 3, and 5 years follow-up
Cardiovascular mortality | 1, 3, and 5 years follow-up

SECONDARY OUTCOMES:
Rate of receiving vascular revascularization | 1, 3, and 5 years follow-up
Readmission rate for vascular reasons | 1, 3, and 5 years follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Cardiology, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang